CLINICAL TRIAL: NCT05000164
Title: Evaluation of Visual Acuity With a Reusable Toric Multifocal Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR-6383
Record Dates: First submitted 2021-08-03; First posted 2021-08-11 (Actual); Results first posted 2023-01-23 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Visual Acuity

STUDY DESIGN:
Masking Description: Subjects will be unaware of the identity of the investigational product to help reduce potential bias
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Market Product (Experimental): Eligible subjects will be dispensed the study lenses in a bilateral fashion and will be in the treatment for approximately 5 weeks.
  Interventions: Device: Bausch + Lomb Ultra® Multifocal for Astigmatism

INTERVENTIONS:
Device: Bausch + Lomb Ultra® Multifocal for Astigmatism — Study Lens

SUMMARY:
The study is a bilateral, single-masked, single-arm, 4-visit dispensing study evaluating the visual performance of the study lenses.

DETAILED DESCRIPTION:
The study is a bilateral, single-masked, single-arm, 4-visit dispensing study evaluating the visual performance of the study lenses.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all of the following criteria to be enrolled in the study:

  1. Read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
  2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
  3. Be at least 40 and not more than 70 years of age at the time of screening.
  4. Own a wearable pair of spectacles if required for their distance vision.
  5. Be an adapted soft contact lens wearer in both eyes (i.e. has worn lenses a minimum of 2 days per week for at least 8 hours per wear day, for the past month).
  6. Be an existing wearer of a presbyopic contact lens correction (e.g., reading spectacles over contact lenses, multifocal or monovision contact lenses, etc.) or respond positively to at least one symptom on the "Presbyopic Symptoms Questionnaire".
  7. Have distance spherical component of refraction in the range of either -1.25 D to -3.75 D or +1.25 to +3.75 D in each eye.
  8. Have refractive cylinder in the range of -0.75 D to -1.75 D in each eye, with their cylinder axis 90°±25°.
  9. Have near ADD power requirement in the range of +0.75 D to +2.50 D in each eye.
  10. Have best corrected distance visual acuity of 20/20-3 or better in each eye.

      Exclusion Criteria:
* The subject must not:

  1. Be currently pregnant or lactating.
  2. Have any active or ongoing ocular or systemic allergies that may interfere with contact lens wear.
  3. Have any active or ongoing systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear. This may include, but not be limited to, diabetes, hyperthyroidism, Sjögren's syndrome, xerophthalmia, acne rosacea, Stevens- Johnson syndrome, and immunosuppressive diseases or any infectious diseases (e.g. hepatitis, tuberculosis).
  4. Use systemic medications that may interfere with contact lens wear or cause blurred vision. See section 9.1 for additional details regarding excluded systemic medications.
  5. Currently use ocular medication with the exception of rewetting drops.
  6. Have any known hypersensitivity or allergic reaction to single use preservative free rewetting drops, sodium fluorescein, or Biotrue® multipurpose solution.
  7. Have any previous, or planned, ocular or intraocular surgery (e.g. radial keratotomy, PRK, LASIK, lid procedures, cataract surgery, retinal surgery, etc.).
  8. Have a history of amblyopia or strabismus.
  9. Have a history of herpetic keratitis.
  10. Have a history of irregular cornea.
  11. Have a history of pathological dry eye.
  12. Have participated in any contact lens or lens care product clinical trial within 14 days prior to study enrollment.
  13. Be an employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician).
  14. Have clinically significant (Grade 2 or greater) corneal edema, corneal vascularization, corneal staining, tarsal abnormalities or bulbar injection, or any other corneal or ocular abnormalities which would contraindicate contact lens wear.
  15. Have entropion, ectropion, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions.
  16. Have any current ocular infection or inflammation.
  17. Have any current ocular abnormality that may interfere with contact lens wear.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2022-01-13 (Actual); Study Completion 2022-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Vision Care, Inc. Clinical Trial, Study Director — Johnson & Johnson Vision Care, Inc.
Locations (9):
- United States (9):
  - Vue Optical Boutique, Jacksonville, Florida
  - Stam & Associates Eye Care, Jacksonville, Florida
  - VRC-East, Jacksonville, Florida
  - Maitland Vision Center, Maitland, Florida
  - The Eyecare Studio, Decatur, Georgia
  - Ctr For Opht and Vision Rsrch At Eye Associates Of New York, Manhattan, New York
  - Sacco Eye Group, Vestal, New York
  - Vision Boutique, Houston, Texas
  - Botetourt Eyecare LLC, Salem, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 75 subjects were enrolled into this study. Of those enrolled, 72 were dispensed a study lens, while 3 subjects failed to meet all eligibility criteria. Of those dispensed, 62 subjects completed, and 10 subjects discontinued from the study.
Groups:
- Samfilcon A: Subjects that were dispensed the study lens.
Period: Overall Study
Arm/Group | Samfilcon A
Started | 72
Completed | 62
Not Completed | 10
Not completed — Adverse Event | 1
Not completed — Unsatisfactory Visual Response due to Test Article | 1
Not completed — Lens Discomfort | 3
Not completed — Withdrew Consent during Study | 2
Not completed — Subject Withdrawn by PI | 2
Not completed — Other Fractured Test Article | 1

BASELINE CHARACTERISTICS:
Population: All subjects dispensed a study lens.
Arm/Group | Samfilcon A
Number analyzed (Participants) | 72
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.4 (8.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 25
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 3
  Black or African American | 10
  Native Hawaiian or Other Pacific Islander | 1
  White | 58
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 72

OUTCOME MEASURES:

1. Primary Outcome: Binocular High Luminance High Contrast logMAR Visual Acuity
Description: Binocular visual acuity was measured on a logMAR (Logarithm of Minimal Angle of Resolution) scale under high luminance high contrast condition. At distance (4 meters), VA is assessed using ETDRS (Early Treatment Diabetic Retinopathy Study) charts; while near (40 cm) and intermediate (64 cm) assessments were made using reduced Guillon-Poling charts. Letter-by-letter results calculated the visual performance score for each chart read. LogMAR scores closer to zero, or below zero, indicate a better visual acuity. A logMAR visual performance score of 0.0 is equivalent to Snellen visual acuity of 20/20.
Time Frame: 4-Week Follow-up
Population: All completed subjects.
Measure: Mean (Standard Deviation); unit: LogMAR
Groups:
- Samfilcon A: All subjects dispensed the study lens.
Arm/Group | Samfilcon A
Number analyzed (Participants) | 62
LogMAR
  Distance (4m) | -0.13 (0.097)
  Intermediate (64cm) | -0.02 (0.115)
  Near (40cm) | 0.09 (0.139)
Statistical Analysis 1: Comparison: Samfilcon A; Distance (4m); Test type: Superiority; Mixed Models Analysis; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; Least-square Mean = -0.12, 95% CI 2-sided [-0.17 to -0.07], Standard Error of Mean 0.020 — The upper limit of each 95% confidence interval was compared to 0.0 logMAR for distance
Statistical Analysis 2: Comparison: Samfilcon A; Intermediate (64cm); Test type: Superiority; Mixed Models Analysis; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; Least-square Mean = -0.01, 95% CI 2-sided [-0.06 to 0.04], Standard Error of Mean 0.022 — The upper limit of each 95% confidence interval was compared to 0.17 logMAR for intermediate
Statistical Analysis 3: Comparison: Samfilcon A; Near (40cm); Test type: Superiority; Mixed Models Analysis; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; Least-square Mean = 0.09, 95% CI 2-sided [0.04 to 0.15], Standard Error of Mean 0.024 — The upper limit of each 95% confidence interval was compared to 0.17 logMAR for near

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study; approximately 1 month per subject.
Groups:
- Samfilcon A: Subjects dispensed the study lens.
Arm/Group | Samfilcon A
All-Cause Mortality (participants affected / at risk) | 0/72
Serious Adverse Events (participants affected / at risk) | 0/72
Other Adverse Events (participants affected / at risk) | 0/72

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-29): https://cdn.clinicaltrials.gov/large-docs/64/NCT05000164/Prot_SAP_001.pdf